CLINICAL TRIAL: NCT06092177
Title: Evaluation of Virtual Reality Distraction on Dental Anxiety in Patients Undergoing Periodontal Surgery
Brief Title: Virtual Reality Distraction in Patients Undergoing Periodontal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ezgi Gürbüz, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03
Record Dates: First submitted 2023-10-15; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-04

CONDITIONS: Virtual Reality; Oral Surgery; Dental Anxiety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The group will include patients who undergo periodontal surgery with virtual reality distraction
  Interventions: Procedure: Periodontal surgery with virtual reality distraction
- Control group (Experimental): The group will include patients who undergo periodontal surgery without virtual reality distraction
  Interventions: Procedure: Periodontal surgery without virtual reality distraction

INTERVENTIONS:
Procedure: Periodontal surgery with virtual reality distraction — Periodontal surgery to improve gingival contour and eliminate inflamed periodontal pockets
  Arms: Test group
Procedure: Periodontal surgery without virtual reality distraction — Periodontal surgery to improve gingival contour and eliminate inflamed periodontal pockets
  Arms: Control group

SUMMARY:
The goal of this randomized controlled clinical trial is to evaluate the effect of virtual reality technology on anxiety and pain levels in patients undergoing periodontal surgery.

Participants will be randomly assigned into test and control groups. While the patients in the test group will undergo periodontal surgery with virtual reality distraction, the patients in the control group without distraction. After treatment, the groups will be compared regarding anxiety and pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18
* Systemically healthy patients
* Need for periodontal surgical treatment in the mandibular anterior region
* Scoring 15 or above on the modified dental anxiety scale

Exclusion Criteria:

* Having a history of seizures or a convulsive disorder
* Balance disorders such as nystagmus, vertigo
* Use of psychotropic drugs
* Getting treatment for anxiety
* Presence of dermatological lesions on the face, especially around the eyes
* A lesion in the eye that will prevent the use of virtual reality glasses
* Systemic disease and medication use that contraindicate periodontal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Anxiety level | Preoperative, immediately postoperative
  Modified dental anxiety scale where higher scores mean a worse outcome and has a minimum value of 5 and a maximum value of 25

SECONDARY OUTCOMES:
Pain level | Preoperative, immediately postoperative
  Visual analog scale where higher scores mean a worse outcome and has a minimum value of 0 and a maximum value of 10
Systolic blood pressure | Preoperative, intraoperative, immediately postoperative
  Blood pressure will be measured by a sphygmomanometer.
Diastolic blood pressure | Preoperative, intraoperative, immediately postoperative
  Blood pressure will be measured by a sphygmomanometer.
Heart rate | Preoperative, intraoperative, immediately postoperative
  The frequency of the heartbeat measured by the number of contractions of the heart per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Gurbuz, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurbuz E, Gurbuz AA. Investigation of the effect of virtual reality distraction in patients undergoing mandibular periodontal surgery: A randomized controlled study. J Esthet Restor Dent. 2024 May;36(5):813-822. doi: 10.1111/jerd.13203. Epub 2024 Feb 5. PMID 38314536